CLINICAL TRIAL: NCT05980962
Title: Anteriorization of the Inferior Oblique Muscle Versus Anteriorization and Resection for Asymmetrical Dissociated Vertical Deviation With Inferior Oblique Muscle Overaction
Brief Title: Inferior Oblique Muscle Anteriorization Versus Anteriorization and Resection in DVD With IOOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ghada Osama Mohamed, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-97-2018
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Dissociated Vertical Deviation; Inferior Oblique Overaction
Keywords: DVD; IOOA; IO Anteriorization; IO Anteriorization with rescetion
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Anteriorization group) (Active Comparator): Symmetrical Anteriorization of the inferior oblique muscle
  Interventions: Procedure: Inferior oblique anteriorization
- Group 2 (Resction group) (Experimental): Asymmetrical Anteriorization of the inferior oblique muscle, where an additional resection of the inferior oblique was done for the eye with the larger deviation
  Interventions: Procedure: Inferior oblique anteriorization together with unliateral resction

INTERVENTIONS:
Procedure: Inferior oblique anteriorization — symmterical anteriorization the the inferior oblique muscle 1 mm behind and lateral to the inferior rectus insertion
  Arms: Group 1 (Anteriorization group)
Procedure: Inferior oblique anteriorization together with unliateral resction — asymmterical surgery, anteriorization the the inferior oblique muscle 1 mm behind and lateral to the inferior rectus insertion in one eye, and an additional 3-5 mm resction of the inferior oblique in the eye with the larger devation
  Arms: Group 2 (Resction group)

SUMMARY:
The goal of this clinical trial is to compare the results of two surgical modalities in patients with Dissociated vertical deviation with inferior oblique muscle overaction . The main questions it aims to answer are:

* How much does the magnitude of DVD improve after each modality?
* Is the IOOA eliminated? Participants will be divided into two equal groups; Researchers will compare the efficacy of symmetrical anteriorization of the inferior oblique and adding an additional rescetion to one eye in the second group to see which group had more signifcant reduction in the magnitude of DVD and IOOA.

DETAILED DESCRIPTION:
A prospective study was performed on patients with bilateral symmterical dissociated vertical deviation(DVD) and bilateral inferior oblique muscle overaction (IOOA) in Cairo University hospitals starting from February 2018 through December 2021. Patients wetre included in the study if they had a minimum follow up period of 6 months. The study included 54 patients (108 eyes) with manifest DVD and IOOA in boths eyes. Patients were divided into two equal groups. The paitents in group 1 underwent symmetrical inferior oblique muscle anteriorization, while the patients in group 2 underwent ayymmetrical surgery , where inferior oblique anteriorization was performed in one eye the same manner is in group 1, and the eye with the larger deviation had an additional 3-5 mm rescetion of the inferior oblique muscle along with anteriorization according to the measured DVD difference between both eyes, whether less than or more than 5 prism diopters respectively.

ELIGIBILITY:
Inclusion Criteria:

* Manifest DVD decompensated to a tropia with free ocular motility
* Cases with or without horizontal misalignment
* Cases with or without previous horizontal muscle surgery

Exclusion Criteria:

* Incomitant, Paralytic or restrictive strabismus
* Eyes with previous inferior oblique muscle surgery
* Recurrent DVD after surgical treatment
* Eyes with previous scleral buckling for retinal deatchment

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
reduction of the magnitude of DVD | 1 week ,1 month, three months, six months
  degree of reduction of the deviation measured in prism diopters

SECONDARY OUTCOMES:
reduction of magnitude of IOOA | 1 week ,1 month, three months, six months
  redctuon in the measured degree of IOOA

CONTACTS AND LOCATIONS:
Overall Officials: Hala M. Elhiliali, Study Chair — Cairo University; Magda S. Abdel-Aziz, Study Director — Cairo University; Heba M. Fouad, Study Director — Cairo University; Ghada O. Mohamed, Principal Investigator — Cairo University
Locations (1):
- Kasr Alainy School of Medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No